CLINICAL TRIAL: NCT04234529
Title: Impact of AMATEA™️ on Physiological Measures and Gaming Performance in Active Gamers: a Placebo Controlled, Double-blind, Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Applied Food Sciences Inc. (Industry)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of School of Health Studies, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO-FY2020-65
Record Dates: First submitted 2019-12-09; First posted 2020-01-21 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Healthy
Keywords: AMATEA; video games; gaming; energy supplement
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Participants will receive each of the 3 interventions over a 3 week period i.e. one acute dose once per week. The 3 interventions include 1) AMATEA, 2) Caffeine, or 3) Placebo
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AMATEA (Active Comparator): 3x 450mg capsules of AMATEA which contains 270mg of caffeine total
  Interventions: Dietary Supplement: AMATEA™
- Caffeine (Active Comparator): 3x 450mg capsules each containing 360mg of microcellulose and 90mg of caffeine (270mg caffeine total)
  Interventions: Dietary Supplement: Caffeine
- Placebo (Placebo Comparator): 3x 450mg capsules of microcellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: AMATEA™ — AMATEA™ is a patented dietary supplement consisting of a unique blend of caffeine and polyphenol antioxidants; standardized at 20% caffeine, 30% chlorogenic acids (similar to green coffee).
  Total of 1.35g of AMATEA containing 270mg of caffeine.
  Arms: AMATEA
Dietary Supplement: Caffeine — 1.08g of microcellulose and 270mg of caffeine.
  Arms: Caffeine
Other: Placebo — 1.35g of microcellulose
  Arms: Placebo

SUMMARY:
AMATEA™ is a patented dietary supplement consisting of a unique blend of caffeine and polyphenol antioxidants; standardized at 20% caffeine, 30% chlorogenic acids (similar to green coffee). In-house evaluations and anecdotal findings related to AMATEA have noted sustained energy without the typical "crash" and/or "jitters" experienced by some with caffeine ingestion alone.

The aim of the present study is to compare the effects of AMATEA and caffeine alone on various measures of cognitive performance, mood, and gaming performance in men and women who regularly engage in gaming activity. The investigators hypothesize that both AMATEA and caffeine will improve outcome measures more than placebo, with greater improvement noted for the AMATEA condition due to the addition of the chlorogenic acid.

DETAILED DESCRIPTION:
The activity of "gaming" is increasing in popularity each year, with millions of young adults engaged in regular play. This has fueled the rise in nutrition and dietary supplementation strategies to aid gaming performance. Since caffeine has been widely used for purposes of improving athletic performance with both relatively low and high dosages, and more recently as a potential aid for "mind" games such as chess at a dosage of 400mg, this has been the nutrient of focus for many gamers. Other multi-component products are making their way to the market.

Active gamers claim to ingest such products regularly throughout their gameplay, which can span from 4-12 hours per session for regular gamers. AMATEA™ is a patented dietary supplement consisting of a unique blend of caffeine and polyphenol antioxidants; standardized at 20% caffeine, 30% chlorogenic acids (similar to green coffee). The product is also Generally Recognized as Safe (GRAS) and USDA organic.

While caffeine has been well-investigated for its performance boosting effects, chlorogenic acid has been reported to offer many potential health benefits. Specifically, it has been reported to improve select cognitive measures following regular intake, which may translate into more efficient performance with complex tasks-such as those involved with gaming.

In-house evaluations and anecdotal findings related to AMATEA have noted sustained energy without the typical "crash" and/or "jitters" experienced by some with caffeine ingestion alone. While caffeine can prove beneficial to many, some users experience "crashing" 2-3 hours post ingestion, while others feel too "wired" following use and may experience difficulty concentrating. AMATEA contains a relatively low concentration of caffeine per capsule (150mg) in an attempt to avoid such problems, while also containing chlorogenic acid. This may aid gamers who need to maintain fine motor skills and those who need to concentrate on complex activities for several hours continuously.

The aim of the present study is to compare the effects of AMATEA and caffeine alone on various measures of cognitive performance, mood, and gaming performance in men and women who regularly engage in gaming activity. The investigators hypothesize that both AMATEA and caffeine will improve outcome measures more than placebo, with greater improvement noted for the AMATEA condition due to the addition of the chlorogenic acid.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40 years
* male or female
* body mass index (BMI) between 18-34.9 kg/m2
* not be using tobacco products
* no diagnosed history of diabetes
* no diagnosed history of cardiovascular disease
* no diagnosed history of neurological disease
* no consumption of alcohol within 48 hours of testing
* consume < 400mg caffeine daily
* no consumption of caffeine-containing beverages within at least 48 hours of testing
* blood metabolic parameters within normal limits
* if female, not be pregnant
* active gamers: playing at least 4 days per week, for at least 4 hours per day, for the past 12 months
* regularly playing the game Fortnite, for the past 3 months
* willing to play on our console systems and use their personal headset

Exclusion Criteria:

* individuals younger than 18 years or greater than 40 years
* individuals weighing less than 115 pounds
* individuals with a BMI less than 18kg/m2 or greater than 35kg/m2
* individuals with a diagnosed history of diabetes, cardiovascular disease, or neurological disease
* individuals that consume greater than 400mg caffeine daily
* pregnant females
* non-active gamers

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Fortnite Gaming metrics with AMATEA | During 4 hours of gaming following AMATEA ingestion
  We will determine the change in the Fortnite gaming metrics report following 4 hours of play when taking AMATEA versus placebo or caffeine
Fortnite Gaming metrics with caffeine | During 4 hours of gaming following caffeine ingestion
  We will determine the change in the Fortnite gaming metrics report following 4 hours of play when taking caffeine versus placebo or AMATEA
Fortnite Gaming metrics with placebo | During 4 hours of gaming following placebo ingestion
  We will determine the change in the Fortnite gaming metrics report following 4 hours of play when taking placebo versus AMATEA or caffeine
Change in mental performance from baseline with AMATEA | Prior to and during the 6 hour period following AMATEA ingestion
  We will determine the change in daily mental performance assessed via AX-CPT when taking AMATEA versus caffeine or placebo
Change in mental performance from baseline with caffeine | Prior to and during the 6 hour period following caffeine ingestion
  We will determine the change in daily mental performance assessed via AX-CPT when taking caffeine versus caffeine or AMATEA
Change in mental performance from baseline with placebo | Prior to and during the 6 hour period following placebo ingestion
  We will determine the change in daily mental performance assessed via AX-CPT when taking placebo versus caffeine or AMATEA
Change in blood cortisol from baseline with AMATEA | Prior to and during the 6 hour period following AMATEA ingestion
  We will determine the change in daily blood cortisol when taking AMATEA versus caffeine or placebo
Change in blood cortisol from baseline with caffeine | Prior to and during the 6 hour period following caffeine ingestion
  We will determine the change in daily blood cortisol when taking caffeine versus AMATEA or placebo
Change in blood cortisol from baseline with placebo | Prior to and during the 6 hour period following placebo ingestion
  We will determine the change in daily blood cortisol when taking placebo versus AMATEA or caffeine
Change in digital symbol substitution from baseline with AMATEA | Prior to and during the 6 hour period following AMATEA ingestion
  We will determine the change in digital symbol substitution when taking AMATEA versus caffeine or placebo
Change in digital symbol substitution from baseline with caffeine | Prior to and during the 6 hour period following caffeine ingestion
  We will determine the change in digital symbol substitution when taking caffeine versus AMATEA or placebo
Change in digital symbol substitution from baseline with placebo | Prior to and during the 6 hour period following placebo ingestion
  We will determine the change in digital symbol substitution when taking placebo versus AMATEA or caffeine
Change in reaction time from baseline with AMATEA | Prior to and during the 6 hour period following AMATEA ingestion
  We will determine the change in reaction time when taking AMATEA versus caffeine or placebo
Change in reaction time from baseline with caffeine | Prior to and during the 6 hour period following caffeine ingestion
  We will determine the change in reaction time when taking caffeine versus AMATEA or placebo
Change in reaction time from baseline with placebo | Prior to and during the 6 hour period following placebo ingestion
  We will determine the change in reaction time when taking placebo versus AMATEA or caffeine

SECONDARY OUTCOMES:
Heart rate | Prior to and during the 6 hour period following supplement/placebo ingestion
  Change in heart rate each hour after ingestion
Blood pressure | Prior to and during the 6 hour period following supplement/placebo ingestion
  Change in blood pressure each hour after ingestion
Rate pressure product | Prior to and during the 6 hour period following supplement/placebo ingestion
  Change in rate pressure product each hour after ingestion
Digital symbol substitution test | Prior to and during the 6 hour period following supplement/placebo ingestion
  Change in digital symbol substitution test each hour after ingestion
Brunel Mood Score | Prior to and during the 6 hour period following supplement/placebo ingestion
  Change in Brunel Mood Score (Brums-32) using a scale 0 (Not at all) to 4 (Extremely) with higher scores indicating stronger feelings each hour after ingestion
Subjective Mood | Prior to and during the 6 hour period following supplement/placebo ingestion
  Change in subjective mood using a visual analog schedule running from None to Extreme, where values nearer extreme indicate stronger feelings each hour after ingestion
Reaction time | Prior to and during the 6 hour period following supplement/placebo ingestion
  Change in reaction time each hour after ingestion
Blood cortisol | Prior to and during the 6 hour period following supplement/placebo ingestion
  Change in blood cortisol from baseline every 2 hours after ingestion for 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, Ph.D., Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided